CLINICAL TRIAL: NCT04676672
Title: NEOS - A Post-market Clinical Follow-up Study in Patients With Acute or Chronic Aortic Dissection or Aortic Aneurysm Treated With E-vita OPEN NEO
Brief Title: A PMCF Study in Patients With Acute or Chronic Aortic Dissection or Aortic Aneurysm Treated With E-vita OPEN NEO
Acronym: NEOS
Status: Active, not recruiting | Type: Observational
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: NEOS
Record Dates: First submitted 2020-12-07; First posted 2020-12-21 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Aortic Dissection; Aortic Aneurysm
Keywords: Thoracic; Aorta; Aneuysm; Dissection; Open; Repair; Frozen; Elephant; Trunk
MeSH Terms: conditions — Aortic Dissection; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Open repair — Open repair of the aortic arch and descending aorta with or without involvment of the ascending aorta using a hybrid graft.

SUMMARY:
The NEOS post-market clinical follow-up study is undertaken to demonstrate the safety and clinical performance of E-vita OPEN NEO in the treatment of aneurysm or dissection in the ascending aorta, aortic arch and descending thoracic aorta.

DETAILED DESCRIPTION:
In this study, patients will be observed who receive an E-vita OPEN NEO implant for the treatment of thoracic aneurysm or acute or chronic thoracic dissection. E-vita OPEN NEO will be implanted according to the instructions for use and at the discretion of the treating physician.

Participating physicians will provide their observations collected during routine care for patients treated with E-vita OPEN NEO. Written informed consent, specifically allowing the use of clinical records for this observational study, will be obtained from every patient prior to data collection.

The period of data collection will be approximately 60 months from the date of intervention for each patient. Source data verification will be performed on 100% of the patients; data from all the visits that was provided in the database will be reviewed and verified against existing source documents. Complete DICOM image files of the CT scans will be sent to the CoreLab for independent evaluation. All adverse events defined prior to study start will be adjudicated by the Clinical Event Committee (CEC).

ELIGIBILITY:
Inclusion Criteria:

* Patient´s age is between 18 and 75 years.
* Patient is willing and able to comply with the standard follow-up visits planned after the implantation procedure.
* Patient is willing and able to give informed consent.
* Patient satisfies one of the following categories:
* Patient has acute / subacute aortic dissection and requires repair or replacement of damaged or diseased vessels of the aortic arch (with or without involvement of the ascending aorta), and the descending aorta requires treatment, or, in the opinion of the investigator, the patient would derive clinical benefit from prophylactic treatment of the descending aorta.
* Patient has chronic aortic dissection which requires repair or replacement of damaged or diseased vessels of the aortic arch and descending aorta with or without involvement of the ascending aorta, and the patient satisfies one or more of the following criteria:

Patient has aortic sinus, or ascending aorta, or aortic arch, or descending aorta diameter ≥ 5.5 cm.

Patient has aorta diameter < 5.5 cm and a growth rate of ≥ 0.5 cm / year. Patient has ascending aorta diameter ≥ 4.5 cm and requires an aortic valve repair or replacement.

Patient has clinical signs of abdominal or peripheral malperfusion.

* Patient has a fusiform or saccular aortic aneurysm which requires repair or replacement of damaged or diseased vessels of the aortic arch and descending aorta with or without involvement of the ascending aorta, and patient satisfies the following criteria:

Patient has a suitable distal sealing area in the descending thoracic aorta proximal to the celiac trunk.

And in case of fusiform aneurysm one of the following characteristics:

Patient has aortic sinus, or ascending aorta, or aortic arch, or descending aorta diameter ≥ 5.5 cm.

Patient has aorta diameter < 5.5 cm and a growth rate of ≥ 0.5 cm / year. Patient has ascending aorta diameter ≥ 4.5 cm and requires an aortic valve repair or replacement.

* Patient is hemodynamically stable without pharmacological support at time of admission to the hospital (stable blood pressure and heart rate, no shock).

Exclusion Criteria:

* Patient is unfit for open surgical repair involving circulatory arrest.
* Patient has known sensitivities or allergies to nitinol, polyester, platinum-iridium, or polyethylene.
* Patient has systemic infection.
* Patient has endocarditis or active infection of the aorta.
* Patient has a free ruptured aorta.
* Patient has acute stroke or suspected acute stroke.
* Patient is on inotropes at time of arrival to the hospital.
* Patient needs mitral valve repair or replacement.
* Patient is enrolled or plans to be enrolled in another active study.
* Patient is pregnant or breastfeeding or planning to become pregnant during the course of the study.
* Patient has uncorrectable bleeding anomaly (i.e., thrombocytopenia).
* Patient has an eGFR < 45 ml/min/1.73m2 before the intervention
* Patient has known sensitivity to radiopaque contrast agents that cannot be adequately pre-treated.
* Patient has co-morbidity (i.e. active malignancy (progressive, stable or partial remission)) causing expected survival to be less than 3 years.
* Patient has any other medical, social or psychological problems, that in the opinion of the investigator, preclude the patient from participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with thoracic aortic dissection or aneurysm who are eligible for surgical treatment with the frozen elephant trunk technique according to the instructions for use for E-vita OPEN NEO and scheduled for implantation of E-vita OPEN NEO at their physician's discretion in accordance with the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30-day
  Rate of all-cause mortality

SECONDARY OUTCOMES:
Mortality | 3-6, 12, 24, 36, 60 months
  Rate of all-cause mortality
Mortality | 30-day, 3-6, 12, 24, 36, 60 months
  Rate of aortic related mortality
Major Adverse Events | 12 months
  Rate of patients who are free from Major Adverse Events (MAEs) (new permanent disabling stroke (mRS ≥ 2 and at baseline mRS < 2), new permanent (> 30 days) paraplegia or paraparesis, reintervention (excluding reoperation for bleeding or planned or unplanned additional intervention), all-cause mortality)
Device technical success | 24 hours
  Rate of patients with device technical success
Procedural success | At discharge, an avarage of 30 days
  Rate of patients with procedural success
Treatment success | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with treatment success
Aortic rupture | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with aortic rupture
Additional intervention | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with planned or unplanned additional intervention
Reintervention | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with reintervention
Disabling stroke | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with new disabling stroke
Paraplegia | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with new permanent (> 30 days) paraplegia
Paraparesis | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with new permanent (> 30 days) paraparesis
Renal failure | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with renal failure requiring permanent (> 90 days) dialysis or hemofiltration in a patient with a normal pre-procedure serum creatinine level
Aortic regurgitation | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with increase in aortic regurgitation grade of greater than 1 compared to pre-operative measurement
Stenosis | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with stenosis in the supra-aortic head vessels (0 - 30 %, >30 % - 50 %, > 50 % - 70%, > 70%)
Patency | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with patent supra-aortic head vessels
Migration | 3-6, 12, 24, 36, 60 months
  Rate of patients with retrograde migration > 10 mm of the distal end of the stented part of E-vita OPEN NEO
Integrity | At discharge, an avarage of 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with failure of integrity of the E-vita OPEN NEO
Endoleak type Ib (aneurysm) | 3-6, 12, 24, 36, 60 months
  Rate of patients with aneurysm that have an endoleak type Ib
Endoleak type II (aneurysm) | 3-6, 12, 24, 36, 60 months
  Rate of patients with aneurysm that have an endoleak type II
Endoleak type III (aneurysm) | 3-6, 12, 24, 36, 60 months
  Rate of patients with aneurysm that have an endoleak type III
Endoleak type IV (aneurysm) | 3-6, 12, 24, 36, 60 months
  Rate of patients with aneurysm that have an endoleak type IV
Increasing aortic diameter | 12, 24, 36, 60 months
  Rate of patients with aneurysm that have an increasing maximum aortic diameter in the stented region (E-vita OPEN NEO) compared to first post-operative CT
Stable aortic diameter | 12, 24, 36, 60 months
  Rate of patients with aneurysm that have a stable maximum aortic diameter in the stented region (E-vita OPEN NEO) compared to first post-operative CT
Decreasing aortic diameter | 12, 24, 36, 60 months
  Rate of patients with aneurysm that have a decreasing maximum aortic diameter in the stented region (E-vita OPEN NEO) compared to first post-operative CT
Endoleak type Ib (dissection) | 3-6, 12, 24, 36, 60 months
  Rate of patients with dissection that have an endoleak type Ib
Endoleak II (dissection) | 3-6, 12, 24, 36, 60 months
  Rate of patients with dissection that have an endoleak type II
Endoleak type R (dissection) | 3-6, 12, 24, 36, 60 months
  Rate of patients with dissection that have an endoleak type R
Increasing or stable true lumen size | 3-6, 12, 24, 36, 60 months
  Rate of patients with increasing (≥ 5 mm) or stable true lumen in the stented region
Stable or decreasing false lumen size | 3-6, 12, 24, 36, 60 months
  Rate of patients with stable or decreasing (≤ - 5 mm) false lumen in the stented region
Obliterated false lumen in stented region | 3-6, 12, 24, 36, 60 months
  Rate of patients with obliterated false lumen in the stented region
Completely thrombosed false lumen in stented region | 3-6, 12, 24, 36, 60 months
  Rate of patients with completely thrombosed false lumen in the stented region
Partially thrombosed false lumen in stented region | 3-6, 12, 24, 36, 60 months
  Rate of patients with partially thrombosed false lumen in the stented region
Patent false lumen in stented region | 3-6, 12, 24, 36, 60 months
  Rate of patients with patent false lumen in the stented region
Obliterated false lumen between stent and celiac trunk | 3-6, 12, 24, 36, 60 months
  Rate of patients with obliterated false lumen between the bottom of the stent and the celiac trunk
Completely thrombosed false lumen between stent and celiac trunk | 3-6, 12, 24, 36, 60 months
  Rate of patients with completely thrombosed false lumen between the bottom of the stent and the celiac trunk
Partially thrombosed false lumen between stent and celiac trunk | 3-6, 12, 24, 36, 60 months
  Rate of patients with partially thrombosed false lumen between the bottom of the stent and the celiac trunk
Patent false lumen between stent and celiac trunk | 3-6, 12, 24, 36, 60 months
  Rate of patients with patent false lumen between the bottom of the stent and the celiac trunk
Obliterated false lumen between celiac trunk and aortic bifurcation | 3-6, 12, 24, 36, 60 months
  Rate of patients with obliterated false lumen between the celiac trunk and the aortic bifurcation
Completely thrombosed false lumen between celiac trunk and aortic bifurcation | 3-6, 12, 24, 36, 60 months
  Rate of patients with completely thrombosed false lumen between the celiac trunk and the aortic bifurcation
Partially thrombosed false lumen between celiac trunk and aortic bifurcation | 3-6, 12, 24, 36, 60 months
  Rate of patients with partially thrombosed false lumen between the celiac trunk and the aortic bifurcation
Patent false lumen between celiac trunk and aortic bifurcation | 3-6, 12, 24, 36, 60 months
  Rate of patients with patent false lumen between the celiac trunk and the aortic bifurcation

CONTACTS AND LOCATIONS:
Overall Officials: Martin Grabenwöger, Prof., Principal Investigator — Klinikum Floridsdorf
Locations (2):
- Klinikum Floridsdorf, Vienna, Austria
- Westdeutsches Herzzentrum WHGZ, Essen, Germany

IPD SHARING:
Plan to Share IPD: No